CLINICAL TRIAL: NCT03081546
Title: Cross-Cultural Use of Performance-Based Functional Assessment in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1954
Record Dates: First submitted 2017-03-07; First posted 2017-03-16 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Mild Cognitive Impairment; Healthy Controls
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild Cognitive Impairment (MCI): Persons with age-related Mild Cognitive Impairment (MCI) according to clinical diagnosis, consistent with Alzheimer's Association (AA) and the National Institute on Aging (NIA) diagnostic criteria.
  Must be concurrently enrolled in the Rocky Mountain Alzheimer's Disease Center Bio-AD study (clinicaltrials.gov identifier: NCT02612376).
- Healthy Controls: Community dwelling controls older than 55 years of age that are concurrently enrolled in the Rocky Mountain Alzheimer's Disease Center Bio-AD study (clinicaltrials.gov identifier: NCT02612376).

SUMMARY:
This study plans to assess the effectiveness of performance-based functional assessments (PBFAs) and cognitive assessments in diagnosing Alzheimer's disease in Hispanic/Latino populations. The information from this study will be analyzed with data from the Rocky Mountain Alzheimer's Disease Center Bio-AD study (NCT02612376).

ELIGIBILITY:
Inclusion Criteria:

* Persons with age-related MCI or AD according to clinical diagnosis, consistent with National Institute on Aging-Alzheimer's Association (NIA-AA) diagnostic criteria
* Community-dwelling controls
* Age > 55 years
* Have been enrolled and completed at least one visit in the Bio-AD study and consent to access their data (the Rocky Mountain Alzheimer's Disease Center Bio-AD study (clinicaltrials.gov identifier: NCT02612376))
* Have capacity to provide consent; capacity will be assessed at the time of consent
* Ability to complete baseline assessments
* Has informant (study partner) available to complete functional interviews/survey measures

Exclusion Criteria:

* Presence of concomitant medical, neurological, or psychiatric illness or condition that in the opinion of the investigators would confound interpretation of study results. These include:
* Korsakoff encephalopathy;
* active substance abuse;
* hepatitis C;
* opportunistic brain infection;
* brain tumor;
* active neoplastic disease (skin tumors other than melanoma are not exclusionary; participants with stable prostate cancer may be included at the discretion of the project director);
* multiple sclerosis;
* history of clinically significant stroke;
* current evidence or history in the past 2 years of

  * focal brain lesion,
  * head injury with loss of consciousness in the past year, or
  * DSM-5 criteria for any major psychiatric disorder, including

    1. psychosis,
    2. uncontrolled major depression,
    3. bipolar disorder,
    4. alcohol or substance abuse;
    5. blindness,
    6. deafness or
    7. any other disability which may prevent the participant from participating or cooperating in the protocol.
* Prisoners
* Any contraindication for MRI

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with Mild Cognitive Impairment and healthy aging adults
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
University of California San Diego (UCSD) Performance-Based Skills Assessment (UPSA) | 30 minutes
  Measure independent functioning in everyday life for controls and individuals with MCI
Medication Management Ability Assessment | 15 minutes
  Measure independent management of medications in controls and individuals with MCI
Lawton iADL (instrumental activities of daily living) scale | 5 minutes
  Measure ability to perform instrumental activities of daily living in controls and individuals with MCI

CONTACTS AND LOCATIONS:
Overall Officials: Louis Medina, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States